CLINICAL TRIAL: NCT02172599
Title: The Influence of Sit-stand Workstations Upon Total Physical Activity: a 12 Month Randomised Controlled Trial
Brief Title: Take A Stand for Workplace Health: A Sit-stand Workstation Project Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brunel University (Other)
Collaborators: Macmillan Canceer Support (Other); Ergotron (Unknown); Public Health England (Other Government)
Responsible Party: Principal Investigator, Jennifer Hall, PhD Researcher, Brunel University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: TSWH; R33134 (Other Grant/Funding Number: Macmillan Cancer Support)
Record Dates: First submitted 2014-06-22; First posted 2014-06-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Physical Activity
Keywords: sit-stand workstation; workplace; multi-component intervention; randomised control trial design; physical activity; sitting; sedentary behaviour; process evaluation; health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- multi-component intervention (Experimental): Sit-stand workstation provision
  The multi-component intervention will align with the World Health Authority's promotion of a healthy workplace model, which emphasises that best-practice workplace health interventions should involve an integrated approach involving organisation and individual level approaches to behaviour change (WHO, 2010). Thus, participants will receive a sit-stand workstation with additional support to use the sit-stand workstation.
  Interventions: Behavioral: Sit-stand workstation provision
- Sit-stand workstation only (Experimental): Sit-stand workstation provision
  Participants in this arm will receive a sit-stand workstation. They will not receive any support to use the sit-stand workstation, except some health and safety advice upon installation.
  Interventions: Behavioral: Sit-stand workstation provision
- Usual practice (seated workstation) (No Intervention): This arm is the control group. They will continue to use their usual seated workstation for the duration of the study.

INTERVENTIONS:
Behavioral: Sit-stand workstation provision — The research compares the effects of a sit-stand workstation only and a multi-component sit-stand workstation intervention including individual and organisation-level approaches, with usual office-based working practice (no sit-stand workstation) over 12 months.
  Other Names: Ergotron: workfit-A, workfit-D
  Arms: Sit-stand workstation only; multi-component intervention

SUMMARY:
The purpose of this study is to examine the contribution of sit-stand workstations to total daily physical activity in a multi-component office-based 12 month intervention.

DETAILED DESCRIPTION:
This study adopts a randomised control trial design and is mixed methods (qualitative and quantitative). The outcome data from the trial is quantitative. Alongside this a qualitative process evaluation will be conducted to inform the intervention, explain trial results and understand the intervention implementation and context (Cathain et al. 2014). Two worksites will participate in this study, in line with COCHRANE recommendations for randomised control trials.

ELIGIBILITY:
Inclusion Criteria:

* Must be a full-time employee on a fixed term contract for at least 18 months at one of the two worksites involved in the study (Macmillan Cancer Support, Public Health England)
* Must engage in primarily desk-based work
* Must have their own desk (i.e. does not hot desk) Must be primarily office based (i.e. not working from home)
* Must have no plans to leave the organisation for an extended period (e.g. holiday > 4 weeks or secondment) or finitely before the anticipated study end date (January 2016)

Exclusion Criteria:

* Have engaged in standing-based desk work in the month prior to the start of the study
* Have been advised against standing by a health professional; or be unable to stand
* Work for the Macmillan Support Line

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Measured 5 times over 13 months, for seven days each time. Time points = baseline, 1-2weeks, 3 months, 6 months and 12 months
  ActivPAL:
  Sitting and standing will be measured objectively using the ActivPAL device. The ActivPAL provides reliable measures of total sitting time and standing time, and number of sit-to-stand transitions per hour (Lyden et al. 2012).
  ActiGraph (GT3X+):
  Physical activity intensity and duration will be measured objectively using the ActiGraph activity monitor.The GT3X reliably classifies physical activity intensity in free-living environments (Ozemek et al. 2014).
  Activity diaries:
  These dairies will be used to assess the type and context of physical activity behaviour. A text reminder will be sent to all participants once daily for the duration of the data collection period. Text message models have shown some success in increasing compliance to research (Armstrong et al. 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hall, BSc, Principal Investigator — Brunel University
Locations (2):
- United Kingdom (2):
  - Public Health England, SKipton House, London
  - Macmillan Cancer Support UK Office, London

REFERENCES:
- [Derived] Hall J, Kay T, McConnell A, Mansfield L. "Why would you want to stand?" an account of the lived experience of employees taking part in a workplace sit-stand desk intervention. BMC Public Health. 2019 Dec 17;19(1):1692. doi: 10.1186/s12889-019-8038-9. PMID 31847821
- [Derived] Hall J, Mansfield L, Kay T, McConnell AK. The effect of a sit-stand workstation intervention on daily sitting, standing and physical activity: protocol for a 12 month workplace randomised control trial. BMC Public Health. 2015 Feb 15;15:152. doi: 10.1186/s12889-015-1506-y. PMID 25879905
- See also: This link provides physical activity information for people affected by cancer — http://www.macmillan.org.uk/Cancerinformation/Livingwithandaftercancer/Physicalactivity/Physicalactivity.aspx
- See also: This link provides advice on returning to work for people affected by cancer — http://www.macmillan.org.uk/Cancerinformation/Livingwithandaftercancer/Workandcancer/Supportforemployees/Workcancer/Goingbacktowork.aspx
- See also: This link illustrates the workstation options that will be utilized in this intervention study — http://www.ergotron.com/Products/Workstations/StandUpDesks/tabid/803/language/en-GB/Default.aspx